CLINICAL TRIAL: NCT01190891
Title: A Manual Physical Therapy Approach Versus Subacromial Corticosteroid Injection for Treatment of Shoulder Impingement Syndrome: a Randomized Clinical Trial
Brief Title: Physical Therapy Versus Steroid Injection for Shoulder Impingement Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Madigan Army Medical Center (U.S. Federal Agency)
Collaborators: University of Puget Sound (Other); Franklin Pierce University (Other)
Responsible Party: Principal Investigator, Dan Rhon, Department Research Director, Madigan Army Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 111411-1
Record Dates: First submitted 2010-06-09; First posted 2010-08-30 (Estimated); Results first posted 2016-04-29 (Estimated); Last update posted 2016-04-29 (Estimated); Status verified 2016-03

CONDITIONS: Shoulder Impingement Syndrome
Keywords: Rotator cuff tendonitis; Shoulder pain; Shoulder impingement
MeSH Terms: conditions — Shoulder Impingement Syndrome; Rotator Cuff Injuries; Shoulder Pain | interventions — Musculoskeletal Manipulations; Manipulation, Osteopathic; Adrenal Cortex Hormones; Steroids

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Manual Physical Therapy (Active Comparator): The orthopaedic manual physical therapy (OMPT) intervention approach used in this study will be based on an impairment model. The physical therapist providing the intervention will address the impairments found in the shoulder joints to include the acromioclavicular joint, glenohumeral joint, and scapular-thoracic joints, and cervical/thoracic spine. Patients will receive procedures tailored to their specific impairments. Procedures will include mobilizations and manipulations of the joint and soft-tissues.
  Interventions: Procedure: Manual Physical Therapy
- Corticosteroid Injection (Subacromial) (Active Comparator): Location: Subacromial space; Syringe: 10mL; Needle: 25 gauge, 1.5 inch; Anesthetic: 6 mL of 1% lidocaine or marcaine; Corticosteroid: 1.0 mL Triamcinolone Acetonide (Kenalog), 40 mg/mL
  Interventions: Procedure: Corticosteroid Injection

INTERVENTIONS:
Procedure: Manual Physical Therapy — Same as arm description
  Other Names: Orthopaedic Manual Physical Therapy; Manual Therapy; Osteopathic Manipulative Therapy; Manipulative Therapy
  Arms: Manual Physical Therapy
Procedure: Corticosteroid Injection — Dose represents a glucocorticoid potency of 400 hydrocortisone equivalents/injection (mg).
  Other Names: Steroid Injection
  Arms: Corticosteroid Injection (Subacromial)

SUMMARY:
The purpose of this study is to evaluate and compare the short and long-term effectiveness of two common interventions, manual physical therapy versus corticosteroid injection, for the treatment of shoulder impingement syndrome.

DETAILED DESCRIPTION:
Dysfunction in the shoulder has been reported to affect up to 33% of the general population and generate up to 5% of all consultations from general practitioners. Shoulder problems have been reported as the second highest musculoskeletal complaint for those seeking care from a physical therapist in a deployed environment. Impingement syndromes occur in nearly anyone who repeatedly or forcefully uses their upper extremity in an elevated position, which is very common in the active duty population, and is often characterized by pain during this motion. Managed improperly, this can lead to disruption in work performance and prolonged disability.

Corticosteroid and analgesic injections are some of the most common procedures for orthopedists, rheumatologists, and general practitioners to use in the management of shoulder pain. Conflicting reports from systematic reviews questions the efficacy of corticosteroid injections over other interventions, including oral non-steroidal anti-inflammatory drugs (NSAIDs). Additionally they are not without potential risk such as infection or deleterious effects of prolonged corticosteroid use to include tissue degeneration reported in animal studies as well as other regions of the human body. Manual physical therapy offers a non-invasive approach with negligible risk in as few as three to six sessions and has been shown to improve strength and function in this patient population.

The purpose of this study is to evaluate and compare the effectiveness of two interventions that are commonly used in the management of shoulder impingement syndrome.

1. Evaluate the effect that a subacromial corticosteroid injection has on a subject's function and pain as measured by the Shoulder Pain and Disability Index (SPADI).
2. Evaluate the effect that manual physical therapy has on a subject's function and pain as measured by the Shoulder Pain and Disability Index (SPADI).
3. Compare the effect sizes of the two different interventions in a patient population with shoulder impingement syndrome.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18-65
* Read, write, and speak English
* Tricare beneficiary and eligible for healthcare at a military treatment facility
* Primary complaint of shoulder pain
* Meets diagnostic criteria for shoulder impingement (mentioned below)

To be included in the study participants are required to have:

1. pain with one of the 2 tests in category I, and
2. pain with one test from either category II or category III. * "pain" is defined as reproduction of the usual pain that the subject experiences that makes up the nature of their complaint.

Category I: Impingement signs

1. Passive overpressure at full shoulder flexion with the scapula stabilized.
2. Passive internal rotation at 90 degrees of shoulder flexion in the scapular plane and in progressive degrees of horizontal adduction.

Category II: Active shoulder abduction Active shoulder abduction Category Ill: resisted break tests

1. Abduction
2. Internal rotation
3. External rotation

Exclusion Criteria:

* History of shoulder injection in last 3 months
* History of shoulder dislocation, subluxation, fracture, adhesive capsulitis of the glenohumeral joint, or cervical/shoulder/upper back surgery
* Full-thickness rotator cuff tears
* Presence of cervical radiculopathy, radiculitis, or referral from cervical spine
* Total baseline SPADI score not less than 20% (to prevent a ceiling effect with treatment)
* Prior OMPT treatment to the involved limb for the current episode of pain
* Military service members pending a medical evaluation board, a physical valuation board, or equivalent discharge process, or in medical hold to determine long term disposition. For non-military personnel, anyone that is pending or undergoing any litigation for their injury.
* Contraindication to receiving a corticosteroid injection (allergies, adverse reactions, history of multiple injections in that area even if not within last 30 days, etc)
* Inability to fill out informed consent form
* Unable to come into the clinic for regular treatment over the course of the following month.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 104 (Actual)
Dates: Start 2010-05; Primary Completion 2013-03 (Actual); Study Completion 2013-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Daniel I Rhon, DPT, DSc, Principal Investigator — Madigan Army Medical Center; Joshua A Cleland, PhD, Study Director — Franklin Pierce University
Locations (1):
- Madigan Army Medical Center, Tacoma, Washington, United States

IPD SHARING:
Plan to Share IPD: Yes
Data sharing can only occur after a Data Sharing Agreement has been approved by the US Defense Health Agency

REFERENCES:
- [Background] Arroll B, Goodyear-Smith F. Corticosteroid injections for painful shoulder: a meta-analysis. Br J Gen Pract. 2005 Mar;55(512):224-8. PMID 15808040
- [Background] Koester MC, Dunn WR, Kuhn JE, Spindler KP. The efficacy of subacromial corticosteroid injection in the treatment of rotator cuff disease: A systematic review. J Am Acad Orthop Surg. 2007 Jan;15(1):3-11. doi: 10.5435/00124635-200701000-00002. PMID 17213378
- [Background] Kromer TO, Tautenhahn UG, de Bie RA, Staal JB, Bastiaenen CH. Effects of physiotherapy in patients with shoulder impingement syndrome: a systematic review of the literature. J Rehabil Med. 2009 Nov;41(11):870-80. doi: 10.2340/16501977-0453. PMID 19841837
- [Background] Desmeules F, Cote CH, Fremont P. Therapeutic exercise and orthopedic manual therapy for impingement syndrome: a systematic review. Clin J Sport Med. 2003 May;13(3):176-82. doi: 10.1097/00042752-200305000-00009. PMID 12792213
- [Background] Camarinos J, Marinko L. Effectiveness of manual physical therapy for painful shoulder conditions: a systematic review. J Man Manip Ther. 2009;17(4):206-15. doi: 10.1179/106698109791352076. PMID 20140151
- [Background] Bang MD, Deyle GD. Comparison of supervised exercise with and without manual physical therapy for patients with shoulder impingement syndrome. J Orthop Sports Phys Ther. 2000 Mar;30(3):126-37. doi: 10.2519/jospt.2000.30.3.126. PMID 10721508
- [Derived] Rhon DI, Boyles RB, Cleland JA. One-year outcome of subacromial corticosteroid injection compared with manual physical therapy for the management of the unilateral shoulder impingement syndrome: a pragmatic randomized trial. Ann Intern Med. 2014 Aug 5;161(3):161-9. doi: 10.7326/M13-2199. PMID 25089860
- [Derived] Rhon DI, Boyles RE, Cleland JA, Brown DL. A manual physical therapy approach versus subacromial corticosteroid injection for treatment of shoulder impingement syndrome: a protocol for a randomised clinical trial. BMJ Open. 2011 Jan 1;1(2):e000137. doi: 10.1136/bmjopen-2011-000137. PMID 22021870

RESULTS

PARTICIPANT FLOW:
Groups:
- Manual Physical Therapy: The orthopaedic manual physical therapy (OMPT) intervention approach used in this study was based on an impairment model. The physical therapist providing the intervention addressed impairments found in the shoulder joints to include the acromioclavicular joint, glenohumeral joint, and scapular-thoracic joints, and cervical/thoracic spine. Patients received procedures tailored to their specific impairments. Procedures included mobilizations and manipulations of the joint and soft-tissues.
  Manual Physical Therapy: Same as arm description
Period: Overall Study
Arm/Group | Manual Physical Therapy | Corticosteroid Injection (Subacromial)
Started | 52 | 52
Completed | 46 | 52
Not Completed | 6 | 0
Not completed — Protocol Violation | 1 | 0
Not completed — Withdrawal by Subject | 5 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Manual Physical Therapy | Corticosteroid Injection (Subacromial) | Total
Number analyzed (Participants) | 46 | 52 | 98
Age, Continuous [Mean (Standard Deviation); unit: years] | 40 (12) | 42 (12) | 41 (12)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17 | 14 | 31
  Male | 29 | 38 | 67
Region of Enrollment [Number; unit: participants]
  United States | 46 | 52 | 98

OUTCOME MEASURES:

1. Primary Outcome: Shoulder Pain and Disability Index
Description: The SPADI is a 100-point, 13 item self-administered questionnaire divided into two subscales (pain and disability), with higher scores indicating greater pain and disability. It is responsive to change and accurately discriminates between patients who are improving or worsening. It has high test-retest reliability and internal consistency. The minimal detectable change (MDC) is 18 and the minimally clinically important difference (MCID) is between 8-13 points. The validity and responsiveness to change of SPADI have been described in physical therapy, as well as primary and secondary care settings.
Time Frame: 1 year
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Manual Physical Therapy | Corticosteroid Injection (Subacromial)
Number analyzed (Participants) | 46 | 52
units on a scale | 21.6 [16.0 to 27.2] | 23.1 [17.7 to 28.6]

2. Secondary Outcome: Global Rating of Change
Description: The GROC questionnaire is an instrument that measures overall changes in the quality of life of the subject. The use of a GROC is a common, feasible, and useful method for assessing outcome, and has been shown to be a valid measurement of change in patient status in other pain populations. A change in score of three rating points has been established as a clinically significant in the patients perception of quality of life. The GROC has 15 possible choices, with 0 being equal to no change and -1 to -7 indicating a negative change and +1 to +7 indicating a positive change.
Time Frame: 1 year
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Manual Physical Therapy | Corticosteroid Injection (Subacromial)
Number analyzed (Participants) | 46 | 52
units on a scale | 3 [2 to 4] | 3 [2 to 4]

ADVERSE EVENTS:
Arm/Group | Manual Physical Therapy | Corticosteroid Injection (Subacromial)
Serious Adverse Events (participants affected / at risk) | 0/46 | 0/52
Other Adverse Events (participants affected / at risk) | 0/46 | 0/52

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes